CLINICAL TRIAL: NCT06302049
Title: Clinical Study Evaluating the Safety and Efficacy of Esomeprazole in Treatment of Non-alcoholic Steatohepatitis: A Randomized Controlled Trial.
Brief Title: Clinical Study Evaluating the Safety and Efficacy of Esomeprazole in Treatment of Non-alcoholic Steatohepatitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Aya Hesham Helmy Eltabbakh, Demonstrator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2024-02-28; First posted 2024-03-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Fatty Liver Disease; Steatohepatitis, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esomeprazole group (Experimental): patients in this arm will receive esomeprazole 20 mg once daily
  Interventions: Drug: Esomeprazole
- Placebo group (Placebo Comparator): patients in this arm will receive placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — esomeprazole 20 mg once daily
  Arms: esomeprazole group
Drug: Placebo — Placebo once daily
  Arms: Placebo group

SUMMARY:
The aim of the study is to test the implication of esomeprazole as a possible potential therapy for patients with NASH through evaluating its effect on ultrasound and fibrosis risk scores, serum levels of liver fibrosis biomarkers (fibronectin 1), insulin resistance, metabolic and inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

Both males and females.

* Diabetic and non-diabetic patients.
* Age >18 years old.
* Overweight and obese patient: Body mass index (BMI) ≥ 25 kg/ m2 but <40 kg/ m2.
* Patients with heartburn, peptic ulcer, gastrointestinal reflux disease, erosive esophagitis, Zollinger-Ellison syndrome and helicobacter pylori infection.
* Patients with established diagnosis of NASH based on liver ultrasonography, mild to moderate elevation in aminotransferase activities (>2 but <5 times upper limit of normal), hepatic steatosis index (HIS) >36, HAIR score of 2 or 3.

Exclusion Criteria:

* Patients with a history of hypersensitivity to esomeprazole.
* Patients with BMI ≥ 40 kg/ m2.
* Patients taking warfarin, clopidogrel, digoxin, diazepam and phenytoin to avoid drug-drug interactions as these drugs are CYP2C19 substrates.
* Patients infected with human immune deficiency virus taking antiretroviral medicines or dosage forms containing rilpivirine.
* Patients with a history of viral hepatitis, autoimmune hepatitis, sclerosing cholangitis, biliary obstruction, primary biliary cirrhosis, hemochromatosis, Wilson's disease and alpha-1 antitrypsin deficiency.
* Patients on medications associated with steatosis such as NSAIDs, amiodarone, tamoxifen, estrogen, sodium valproate, corticosteroids, and methotrexate.
* Patients with cancer or with a history of cancer.
* Patients with cardiovascular diseases.
* Pregnant and lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in non-alcoholic fatty liver disease (NAFLD) fibrosis score (NFS) | Before and after 3 months of the intervention
  Increase in NAFLD fibrosis score indicates high probability of advanced liver fibrosis Score lower than -1.5 indicates low probability of advanced liver fibrosis (F0-F2).
  Score higher than or equals -1.5 to < 0.67 indicates intermediate probability of advanced liver fibrosis.
  Score higher than or equals 0.67 indicates high probability of advanced liver fibrosis (F3-F4)

SECONDARY OUTCOMES:
Liver function improvement | Before and after 3 months of the intervention
  change in the other measured parameters such as liver panel
Reduction of oxidative stress | Before and after 3 months of the intervention
  Decrease in the serum level of malondialdehyde (MDA)

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be supplied upon a reasonable request